CLINICAL TRIAL: NCT00595920
Title: An Open-Label Extension Study to Evaluate the Safety, Tolerability and Efficacy of Subcutaneous Tovaxin in Subjects Previously Treated in the TERMS Study 2005-00
Brief Title: Open Label Extension of Prior TERMS Study to Treat Relapsing Forms of Multiple Sclerosis
Acronym: OLTERMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Financial Constraints
Sponsor: Opexa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-00
Record Dates: First submitted 2008-01-03; First posted 2008-01-16 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Clinically Isolated Syndrome
Keywords: Tovaxin; Autologous; T-cell vaccine (TCV)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — tovaxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tovaxin, open-label (Experimental): Tovaxin; 30-45 million autologous myelin reactive T cells
  Interventions: Biological: Tovaxin

INTERVENTIONS:
Biological: Tovaxin — 2 mL subcutaneous injections administered by a healthcare provider at weeks 0, 4, 8, 12, and 24 every year as required.
  Other Names: Autologous TCV; T Cell Vaccine

SUMMARY:
The purpose of this study is to further evaluate the safety and efficacy of Tovaxin in the treatment of relapsing forms of multiple sclerosis.

DETAILED DESCRIPTION:
The subjects with positive myelin-reactive T cells (MRTC) in their blood during the previous TERMS study will immediately be eligible for Tovaxin production and treatment in this open label extension study. The MRTC negative subjects will be monitored quarterly for safety, MRTC reactivity, paraclinical and clinical effect. Subjects who become MRTC positive during the monitoring phase will then be eligible for Tovaxin production and treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the TERMS study and received at least 1 study treatment injection
* Signed and dated statement of informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Experienced a serious adverse drug reaction with confirmatory relationship to Tovaxin in the TERMS study.
* Withdrew from TERMS study and did not continue participating in the remaining 52-week core TERMS study assessments.
* Non-compliant with TERMS study.
* Diagnosis of progressive-relapsing, secondary progressive or primary progressive Multiple Sclerosis (MS) while enrolled in the TERMS study.
* Medical, psychiatric or other conditions that compromise the subject's ability to give informed consent, to understand the patient information, to comply with the study protocol, or to complete the study.
* Any significant change in the subject's medical condition after enrollment in the TERMS study which would have lead to his/her exclusion from participation in that study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Fox, MD, PhD, Principal Investigator — Central Texas Neurology Consultants
Locations (27):
- United States (27):
  - North Central Neurology Associates, PC, Cullman, Alabama
  - Xenoscience - 21st Century Neurology, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Alta Bates Summit Medical Center - East Bay Physicians Medical Group, Berkeley, California
  - Patricia A Fodor, PC, Colorado Springs, Colorado
  - Bradenton Neurology, Bradenton, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Medical College of Georgia - Department of Neurology, Augusta, Georgia
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Allied Physicians Inc, Fort Wayne, Indiana
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, Lexington, Kentucky
  - St Mary's of Michigan - Field Neuroscience Institute, Saginaw, Michigan
  - Ayres & Associates Clinical Trials, Lebanon, New Hampshire
  - Upstate Clinical Research, LLC, Albany, New York
  - Winthrop University Hospital - Clinical Trials Unit, Mineola, New York
  - Neurology Consultants of the Carolinas, PA, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Neurological Research Institute, Columbus, Ohio
  - Neurology Specialists, Inc, Dayton, Ohio
  - Providence St. Vincent Medical Center - Northwest MS Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Maxine Mesinger MS Clinic/Baylor College of Medicine, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - MS Center at Evergreen, Kirkland, Washington

REFERENCES:
- [Background] Zhang J. T-cell vaccination in multiple sclerosis: immunoregulatory mechanism and prospects for therapy. Crit Rev Immunol. 2001;21(1-3):41-55. PMID 11642613
- [Background] Zhang JZ, Rivera VM, Tejada-Simon MV, Yang D, Hong J, Li S, Haykal H, Killian J, Zang YC. T cell vaccination in multiple sclerosis: results of a preliminary study. J Neurol. 2002 Feb;249(2):212-8. doi: 10.1007/pl00007867. PMID 11985389
- [Background] Zhang J. T-cell vaccination for autoimmune diseases: immunologic lessons and clinical experience in multiple sclerosis. Expert Rev Vaccines. 2002 Oct;1(3):285-92. doi: 10.1586/14760584.1.3.285. PMID 12901569

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Extension: 30-45 million autologous myelin reactive T cells
  Tovaxin: 2 mL subcutaneous injections administered by a healthcare provider at weeks 0, 4, 8, 12, and 24 every year as required.
Period: Overall Study
Arm/Group | Open Label Extension
Started | 116
Patients Dosed | 38 (116 patients enrolled; however, only 38 received at least 1 dose.)
Completed | 0
Not Completed | 116
Not completed — The OLTERMS study was discontinued by th | 116

BASELINE CHARACTERISTICS:
Population: Randomized and received at least one dose.
Arm/Group | Open Label Extension
Number analyzed (Participants) | 38
Age, Continuous [Mean (Full Range); unit: years] | 39.98 [21 to 57]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Changes in Number of Combined Unique Active Lesions on Brain Magnetic Resonance Imaging (MRI)
Description: This extension study was discontinued due to financial constraints of the company. Of the 38 patients dosed, 32 did not complete all 5 doses. Of the 6 patients that completed the 5 doses, 5 patients did not have a Wk 52 MRI and therefore, no efficacy results are summarized as there is no comparison data.
Time Frame: Annually
Population: This extension study was discontinued due to financial constraints. No efficacy results are summarized due to the small number of patients who received full treatment and follow-up.
Arm/Group | Open Label Extension
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate Changes in Rate and Severity of Multiple Sclerosis (MS) Progression
Time Frame: Annually
Reporting Status: Not Posted

3. Secondary Outcome: Evaluate Changes in Annualized Relapse Rate
Time Frame: Annually
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Open Label Extension
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Extension (N=38)
Multiple Sclerosis Relapse (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Extension (N=38)
Injection site reaction-Bruising (General disorders) | 11 (11)
Injection site reaction-Disomfort (General disorders) | 7 (7)
Injection site reaction-Induration (General disorders) | 5 (5)
Injection site reaction-Redness (General disorders) | 24 (24)
Injection site reaction-Swelling (Gastrointestinal disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days